CLINICAL TRIAL: NCT01111045
Title: A Phase 2, Double Blind, Randomized, Placebo-Controlled, Proof of Concept, Dose Finding Study of Intraarticular Bone Morphogenetic Protein (BMP-7) in Subjects With Osteoarthritis (OA) of the Knee
Brief Title: Dose Finding Study of Bone Morphogenetic Protein 7 (BMP-7) in Subjects With Osteoarthritis (OA) of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stryker Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09-OA-002
Record Dates: First submitted 2010-04-23; First posted 2010-04-27 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Bone Morphogenetic Protein 7

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 (Active Comparator): 0.03 mg/ml BMP-7, single intraarticular knee injection
  Interventions: Drug: Bone morphogenetic protein 7
- Arm 2 (Active Comparator): 0.1 mg/ml BMP-7, single intraarticular knee injection
  Interventions: Drug: Bone morphogenetic protein 7
- Arm 3 (Active Comparator): 0.3 mg/ml BMP-7, single intraarticular knee injection
  Interventions: Drug: Bone morphogenetic protein 7
- Arm 4 (Placebo Comparator): 1 ml placebo, single intraarticular knee injection (control)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bone morphogenetic protein 7 — Comparison of different doses of the drug via single intraarticular knee injection
  Arms: Arm 1; Arm 2; Arm 3
Drug: Placebo — Placebo
  Arms: Arm 4

SUMMARY:
The objectives of the study are to evaluate the safety and efficacy of intraarticular BMP-7 for the treatment of osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory with a diagnosis of OA of the knee with symptoms for at least 6 months and pain on the majority of days in the last 30 days. Symptoms must include knee joint pain.
* A male or female adult age >40 years
* female subjects of childbearing potential must have a negative serum pregnancy test during screening and a negative urine pregnancy test on the day of injection
* Radiographic evidence of at least one tibiofemoral osteophyte and Osteoarthritis Research Society International (OARSI) Atlas joint space narrowing grade of 1 or 2 in the index knee
* WOMAC pain score of >8 at screening and baseline
* Able to comply with the study and give informed consent
* Able to read, write and understand English

Exclusion Criteria:

* A requirement for treatment with opioids for pain relief.
* Unwilling to abstain from NSAIDs and/or other analgesic medications for 48 hours and acetaminophen for 24 hours prior to pain assessments during the study. Subjects taking low dose aspirin for cardiovascular health may remain on their stable dose throughout the study.
* Using a handicap assistance device (i.e., cane, walker) >50% of the time.
* Undergoing new physical therapy or participating in a weight loss or exercise program that has not been stable for at least 3 months prior to screening visit 1 and will not remain stable during their participation in the study.
* History of arthroscopic or open surgery to the index knee in the past 12 months or planned surgery during study.
* History of joint replacement surgery (index knee).
* Received corticosteroid, short acting hyaluronic acid, or other intraarticular injections of the index knee within 3 months of screening and/or not willing to abstain from treatments for the duration of the study
* Received long acting hyaluronic acid injection of the index knee within 6 months of screening and/or not willing to abstain from treatments for the duration of the study.
* History in the past 10 years of reactive arthritis, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, arthritis associated with inflammatory bowel disease, sarcoidosis, amyloidosis or fibromyalgia.
* Clinical signs and symptoms of active knee infection or radiographic evidence of crystal disease other than chondrocalcinosis (i.e., gout and CPPD).
* A history of abnormal laboratory results ≥2.5 x ULN indicative of any significant medical disease, which in the opinion of the investigator, would preclude the subjects participation in the study
* Any of the following abnormal laboratory results during screening:

  1. ALT and AST ≥2.5x ULN
  2. Hemoglobin <11.5 g/dL (Female) or <13.2 g/dL (Male)
  3. WBC <3500 cells/mm3
  4. Lymphocyte count ≤1000 cells/mm3
  5. Serum creatinine ≥1.5 x ULN
  6. Platelet count below the central laboratory lower limit of normal.
* History of malignancy in the past ten years (<10 years), with the exception of resected basal cell, squamous cell of the skin, resected cervical atypia or carcinoma in situ.
* Significant hip pain, ipsilateral to the index knee that may interfere with assessments of index knee pain
* Skin breakdown at the knee where the injection would take place
* A known or clinically suspected infection with human immunodeficiency virus (HIV), or hepatitis C or B viruses
* Participated within 3 months or will participate concurrently in another investigational drug or vaccine study
* A history of drug or alcohol dependence or abuse in the past 3 years
* Previous treatment with BMP-7 or any bone morphogenetic protein
* A female with reproductive capability who is unwilling to use birth control for the duration of the study and/or intends to conceive within 12 months of dosing.
* Other serious, non-malignant, significant, acute or chronic medical or psychiatric illness that, in the judgment of the investigator, could compromise subject safety, limit the subject's ability to complete the study, and/or compromise the objectives of the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2010-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Western Ontario and McMaster Osteoarthritis Index (WOMAC) pain subscale. | Baseline, and at 24 weeks

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Arizona Arthritis and Rheumatology Research, Glendale, Arizona
  - University of Arizona Arthritis Center, Tucson, Arizona
  - Stanford University School of Medicine, Palo Alto, California
  - UC Davis Medical Center, Center for Aging, Sacramento, California
  - Robin Dore, MD, Inc, Tustin, California
  - Boulder Medical Center, PC, Boulder, Colorado
  - Rheumatology Associates of S. Florida, Boca Raton, Florida
  - The Arthritis Center, Palm Harbor, Florida
  - Rheumatology Associates, Stuart, Florida
  - Northwestern Center for Clinical Research, Chicago, Illinois
  - Apex Medical Research, AMR, Inc, Chicago, Illinois
  - Illinois Bone and Joint Institute, Morton Grove, Illinois
  - Johns Hopkins Medical Center, Baltimore, Maryland
  - Klein & Associates, MD, PA, Cumberland, Maryland
  - Arthritis and Osteoporosis Center of Maryland, Frederick, Maryland
  - The Center for Pharmaceutical Research, PC, Kansas City, Missouri
  - Billings Clinic, Billings, Montana
  - The Ohio State University Medical Center, Columbus, Ohio
  - David R. Mandel, MD, Inc., Mayfield Village, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Clinical Research Center of Reading, West Reading, Pennsylvania
  - Baylor Research Institute, Dallas, Texas
  - Houston Institute for Clinical Research, Houston, Texas
  - Houston Medical Research Associates, Houston, Texas
  - Tacoma Center for Arthritis Research, Tacoma, Washington